CLINICAL TRIAL: NCT06626334
Title: Blue Light as an Anti-inflammatory and Analgesic Strategy in Thoracic Trauma: A Randomized Controlled Trial in Adults With Rib Fractures
Brief Title: Blue Light as an Anti-inflammatory and Analgesic Strategy in Thoracic Trauma
Acronym: BLAASTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca E Kotcher, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); Department of Anesthesiology & Perioperative Medicine, University of Pittsburgh (Unknown); Clinical and Translational Science Institute (CTSI), University of Pittsburgh (Unknown)
Responsible Party: Sponsor-Investigator, Rebecca E Kotcher, MD, T32 Postdoctoral Scholar, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24040163; T32GM075770 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Rib Fractures; Pain, Acute
Keywords: Light Therapy; Blue Light Therapy; Pain Control; Analgesia; Immunomodulation; Bright Light Therapy
MeSH Terms: conditions — Rib Fractures; Acute Pain; Agnosia | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Eligible participants who provide informed consent will be randomized 1:1:1 to bright blue light intervention, bright full-spectrum (white) light comparison, and usual light control arms. Permuted block randomization with random block sizes and stratified by age (less than 65 years, greater than or equal to 65 years) will be used for allocation to the three study arms. Assigned lighting interventions will be administered using commercially-available light therapy lamps (Day*Light Classic Plus) fitted with appropriate filters (LEE Filters) and mounted on stands with rolling casters to facilitate bedside use.
Masking Description: This trial is unblinded due to the nature of a lighting intervention, in which participants and investigators will know which intervention is being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Bright Blue Light (Experimental): The light therapy lamp will be covered with a filter selecting for short wavelength blue light (peak 442 nm, intensity ~1400 lux).
  Interventions: Device: Bright Blue Light; Device: Usual Ambient Light
- Bright Full-Spectrum (White) Light (Active Comparator): The light therapy lamp will be covered with a filter modifying only the light's intensity (~1400 lux).
  Interventions: Device: Bright Full-Spectrum (White) Light; Device: Usual Ambient Light
- Usual Ambient Light (Other): Participants assigned to the usual light arm will be exposed only to the usual lighting conditions of the hospital ward.
  Interventions: Device: Usual Ambient Light

INTERVENTIONS:
Device: Bright Blue Light — Bright blue light will be administered using a Day-Light Classic Plus Light Therapy Lamp fitted with a LEE filter (#132, Medium Blue) and mounted on a healthcare-grade stand with rolling casters (Maclocks Rise Freedom Extended). The light intervention will be administered at bedside for 4 hours daily during the morning/early afternoon hours, repeated for up to 3 days.
  Other Names: Carex Day-Light Classic Plus Light Therapy Lamp; CCFDL93011; LEE Filters
  Arms: Bright Blue Light
Device: Bright Full-Spectrum (White) Light — Bright full-spectrum (white) light will be administered using a Day-Light Classic Plus Light Therapy Lamp fitted with a LEE filter (#211 0.9 ND) and mounted on a healthcare-grade stand with rolling casters (Maclocks Rise Freedom Extended). The light intervention will be administered at bedside for 4 hours daily during the morning/early afternoon hours, repeated for up to 3 days.
  Other Names: Carex Day-Light Classic Plus Light Therapy Lamp; CCFDL93011; LEE Filters
  Arms: Bright Full-Spectrum (White) Light
Device: Usual Ambient Light — Across all arms, the usual ambient light in the inpatient room will not be modified.
  For the Bright Blue Light and Bright Full-Spectrum (White) Light arms, light will be added to the environment using a Day-Light Classic Plus Light Therapy Lamp as specified in the corresponding intervention descriptions.
  For the Usual Ambient Light arm, a Day-Light Classic Plus Light Therapy Lamp mounted on a healthcare-grade stand with rolling casters (Maclocks Rise Freedom Extended) will be positioned at a 12-14 inches from eye level with the on/off switch in the off position. The lamp will be positioned in this manner for 4 hours daily during the morning/early afternoon hours, for up to 3 days.
  Other Names: Carex Day-Light Classic Plus Light Therapy Lamp; CCFDL93011

SUMMARY:
The main goal of this clinical trial is to learn if light therapy improves pain and inflammation in adults with painful rib fractures. The main question it aims to answer is:

- Does bright blue light therapy in addition to standard pain treatments improve pain with breathing in adults with painful rib fractures?

Researchers will compare participants who receive bright blue light therapy to participants who receive white light therapy and participants who receive only usual lighting conditions to look for differences in their pain control. In addition to their assigned light treatment, all participants will receive standard pain control treatments.

Participants will be assigned randomly to one of three groups: one-third will be assigned to bright blue light therapy, one-third will be assigned to bright white light therapy, and one-third will be assigned to usual light only. They will receive their assigned light treatment for 4 hours during the morning/early afternoon for up to 3 days while they are in the hospital. On each day they receive the light treatment and on the day after their final light treatment:

* They will be asked twice to rate their pain at rest and with taking a deep breath.
* They will be tested to confirm that they are not experiencing delirium, or confusion related to being in the hospital.
* They will be asked to wear a heart monitor to look for changes in their heart rate.
* Blood samples will be collected to look for changes in inflammation and the circadian clock, the body's natural 24-hour cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Admitted to a single large academic level I trauma center (Presbyterian/Montefiore hospital) within the first 48 hours of traumatic injury
* Greater than or equal to 1 acute rib fracture
* Pain related to rib fracture(s), by one or more of the following criteria: 1. Pain >/= 4/10 at rest, 2. Pain >/= 4/10 with incentive spirometer (IS) use, and/or 3. Inspiratory volume < 1000 cc
* Anticipated length of stay greater than or equal to 48 hours
* Alert, with capacity to provide informed consent

Exclusion Criteria:

* Mechanical ventilation* or non-invasive positive pressure ventilation administered for respiratory insufficiency prior to the time of informed consent
* Delirium (positive CAM screening) at the time of informed consent
* Ocular trauma, which may interfere with the mechanism of action
* Traumatic brain injury (TBI) or history of TBI or stroke, which may interfere with the mechanism of action
* Splenectomy upon admission or history of splenectomy, which may interfere with the mechanism of action
* History of significant ocular dysfunction** (i.e., macular degeneration, glaucoma, cataracts), which may interfere with the mechanism of action
* History of cataract surgery, due to the possibility of blue light filtering intraocular lens placement
* History of bipolar disorder or schizophrenia, which could increase the risk of an adverse reaction to light exposure (i.e., acute mania)
* History of dementia, which would compromise the reliability of pain intensity and delirium measures

  * Or other condition in which a patient cannot open eyes to receive light intervention or report a pain score **Myopia, hyperopia, and/or astigmatism corrected for with contact lenses or spectacle corrective eyeglasses will NOT be a criterion for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Chest wall pain intensity, with incentive spirometer use | Up to 72 hours (assessed twice daily)
  Chest wall pain intensity with deep breathing will be measured using the Numerical Rating Scale, elicited when the participant is taking a full tidal volume breath using their incentive spirometer. The Numerical Rating Scale is an 11-point scale ranging from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable. The scale will then be assessed at multiple timepoints during the 72 hour period of active study participation including twice daily on up to three intervention days (study days 1-3) and once on the morning following the final intervention day (study day 4 or day of discharge). Pain scale values over time will be compared across study arms.

SECONDARY OUTCOMES:
Intensive care unit-free days | 30 days
  Intensive care unit-free days at 30 days is calculated as 30 minus the number of days spent in an intensive care unit. Participants with death occurring within 30 days of enrollment will be assigned 0 ICU-free days. This will be assessed at 30 days using chart review and, for patients discharged from the hospital, confirmed during a single follow-up phone call. Thus, the range for each participant will be from 0 to 30 days. Differences in ICU-free days will be compared across study arms.
Rev-Erb alpha expression | Up to 72 hours (blood samples collected daily)
  Rev-Erb alpha is a circadian clock protein that will be used as a surrogate for circadian clock activation. Rev-Erb alpha expression will be quantified using Western Blot on blood samples collected each morning for up to 4 collections over the course of active study participation. Rev-erb alpha expression over time will be compared across study arms.
IL-6 concentration | Up to 72 hours (blood samples collected daily)
  Pro-inflammatory cytokine IL-6 concentration (pg/mL) will be quantified using ELISA testing on blood samples collected each morning for up to 4 collections over the course of active study participation. IL-6 concentration over time will be compared across study arms.
TNF-alpha concentration | Up to 72 hours (blood samples collected daily)
  Pro-inflammatory cytokine TNF-alpha concentration (pg/mL) will be quantified using ELISA testing on blood samples collected each morning for up to 4 collections over the course of active study participation. TNF-alpha concentration over time will be compared across study arms.
IL-10 concentration | Up to 72 hours (blood samples collected daily)
  Anti-inflammatory cytokine IL-10 concentration (pg/mL) will be quantified using ELISA testing on blood samples collected each morning for up to 4 collections over the course of active study participation. IL-10 concentration over time will be compared across study arms.
Opioid requirements | Up to 72 hours (calculated daily)
  Daily opioid requirements as quantified by standardized oral morphine equivalents (OME) will be calculated daily during up to 72 hours of active study participation using opioid use data abstracted from the electronic medical record and a comprehensive OME conversion table. Opioid requirements over time will be compared across study arms.
Chest wall pain intensity, at rest | Up to 72 hours (assessed twice daily)
  Chest wall pain intensity at rest will be measured using the Numerical Rating Scale, elicited when the participant is at rest. The Numerical Rating Scale is an 11-point scale ranging from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable. The scale will assessed at baseline for the purpose of eligibility screening. The scale will then be assessed at multiple timepoints during the 72 hour period of active study participation, including twice daily during up to three intervention days and once on the morning following the final intervention day. Pain scale values over time will be compared across study arms.
Hospital-free days | 30 days
  Hospital-free days at 30 days is calculated as 30 minus the number of days spent in an acute-care hospital, long-term acute care hospital (LTACH), or in an emergency department (ED). Participants with death occurring within 30 days of enrollment will be assigned 0 hospital-free days. This will be assessed at 30 days using chart review and, for patients discharged from the hospital, confirmed during a single follow-up phone call. Thus, the range for each participant will be from 0 to 30 days. Differences in hospital-free days will be compared across study arms.
Incidence of in-hospital delirium | At 72 hours or date of discharge (assessed daily)
  The presence or absence of delirium will be assessed using the 3-minute diagnostic interview for Confusion Assessment Method-defined delirium (3D-CAM). Based on the bedside assessment, a published algorithm deems the participant either positive or negative for delirium. The assessment will then be administered at multiple timepoints during the 72 hour period of active study participation, including daily on each intervention day (study days 1-3) and on the morning following the final intervention day (study day 4 or day of discharge). The incidence of delirium within this timeframe will be compared across study arms.
Incidence of pulmonary complications | 30 days
  Pulmonary complications are defined by a composite outcome (clinical pneumonia OR respiratory insufficiency requiring non-invasive positive pressure ventilation OR respiratory failure requiring mechanical ventilation). This dichotomous (yes/no) outcome will be assessed for each participant by electronic medical record review at 30 days post-enrollment. The incidence of pulmonary complications within this timeframe will be compared across study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Kotcher, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Presbyterian Hospital, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data may be provided to researchers at the University of Pittsburgh, other institutions and/or federal repositories for the purposes of research collaboration. Sharing will be completed under an approved sharing agreement. In addition to de-identified study data, the Study Protocol, Statistical Analysis Plan, and Analytic Code will be made available to those researchers with an approved sharing agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available beginning 12 months and ending 36 months following article publication. Data will be available to those requesting the data for 1 year after proposal approval.
Access Criteria: Data will be shared with those researchers who provide a methodologically sound proposal. Only those data necessary to achieve the aims in the approved proposal will be shared. De-identified study data as well as the Study Protocol, Statistical Analysis Plan, and Analytic Code will be made available as appropriate. Proposals should be directed to the corresponding author (kotcherre@upmc.edu) and will undergo approval by the study team.

REFERENCES:
- [Background] Marcantonio ER, Ngo LH, O'Connor M, Jones RN, Crane PK, Metzger ED, Inouye SK. 3D-CAM: derivation and validation of a 3-minute diagnostic interview for CAM-defined delirium: a cross-sectional diagnostic test study. Ann Intern Med. 2014 Oct 21;161(8):554-61. doi: 10.7326/M14-0865. PMID 25329203
- [Background] Auriemma CL, Taylor SP, Harhay MO, Courtright KR, Halpern SD. Hospital-Free Days: A Pragmatic and Patient-centered Outcome for Trials among Critically and Seriously Ill Patients. Am J Respir Crit Care Med. 2021 Oct 15;204(8):902-909. doi: 10.1164/rccm.202104-1063PP. No abstract available. PMID 34319848
- [Background] Nielsen S, Degenhardt L, Hoban B, Gisev N. A synthesis of oral morphine equivalents (OME) for opioid utilisation studies. Pharmacoepidemiol Drug Saf. 2016 Jun;25(6):733-7. doi: 10.1002/pds.3945. Epub 2015 Dec 22. PMID 26693665
- [Background] Yuan D, Collage RD, Huang H, Zhang X, Kautza BC, Lewis AJ, Zuckerbraun BS, Tsung A, Angus DC, Rosengart MR. Blue light reduces organ injury from ischemia and reperfusion. Proc Natl Acad Sci U S A. 2016 May 10;113(19):5239-44. doi: 10.1073/pnas.1515296113. Epub 2016 Apr 25. PMID 27114521
- [Background] Lewis AJ, Zhang X, Griepentrog JE, Yuan D, Collage RD, Waltz PK, Angus DC, Zuckerbraun BS, Rosengart MR. Blue Light Enhances Bacterial Clearance and Reduces Organ Injury During Sepsis. Crit Care Med. 2018 Aug;46(8):e779-e787. doi: 10.1097/CCM.0000000000003190. PMID 29727369
- [Background] Griepentrog JE, Zhang X, Lewis AJ, Gianfrate G, Labiner HE, Zou B, Xiong Z, Lee JS, Rosengart MR. Frontline Science: Rev-Erbalpha links blue light with enhanced bacterial clearance and improved survival in murine Klebsiella pneumoniae pneumonia. J Leukoc Biol. 2020 Jan;107(1):11-25. doi: 10.1002/JLB.4HI0519-155R. Epub 2019 Aug 4. PMID 31379019
- [Derived] Kotcher RE, Rosengart MR, La Colla L, Lin HS, Vogt KM, Xu Y, Neal MD. Blue Light as an Anti-inflammatory and Analgesic Strategy in Thoracic Trauma (BLAASTT): protocol for a randomised controlled trial in adult trauma inpatients with painful rib fractures. BMJ Open. 2025 Sep 5;15(9):e097462. doi: 10.1136/bmjopen-2024-097462. PMID 40912706
- See also: Carex Day-Light Classic Plus Light Therapy Lamp — https://carex.com/products/carex-day-light-classic-plus-light-therapy-sun-lamp?gad_source=1&gclid=CjwKCAjw_Na1BhAlEiwAM-dm7A-EDRVyYIrJSjTxxQgV6JfFnyuoSDCshBUMFcD5iV8XU2MIbgSgMRoCYaoQAvD_BwE
- See also: LEE Filter #132 — https://leefilters.com/colour/132-medium-blue/
- See also: LEE Filter #211 0.9ND — https://leefilters.com/colour/211-0-9nd/
- See also: Maclocks Rise Freedom Extended Rolling Kiosk — https://www.maclocks.com/rise-freedom-extended-rolling-kiosk.html